CLINICAL TRIAL: NCT04292470
Title: Physiology of GERD and Treatment Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1485210; K23AT009218 (NIH)
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Results first posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Amitriptyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amitriptyline (Experimental): Amitriptyline 10 mg daily
  Interventions: Drug: Amitriptyline

INTERVENTIONS:
Drug: Amitriptyline — Amitriptyline tablet

SUMMARY:
This study is designed to assess the physiologic and behavioral mechanisms associated with enhanced medication effects in adult patients with functional GERD-related symptoms.

DETAILED DESCRIPTION:
Subjects will complete questionnaires regarding their GERD-related symptoms and have a visit with a study clinician regarding their symptoms. Heart rate variability and galvanic skin response will be measured in the patient-provider dyads and the visits video recorded. Subjects will receive a two-month supply of amitriptyline (10 mg/day), along with instructions for taking it. Subjects will complete a daily GERD symptom diary during the first and eighth weeks of the study. At the end of the 8-week observation period, subjects will complete follow-up measures of GERD symptom severity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 24-64 years old
* Functional heartburn (defined as <4% of time with reflux on 24 hour pH manometry) symptoms 3 or more days per week with an average daily symptom severity of 3 or more on a 7-day baseline symptom diary
* English language proficiency
* Willingness to be videotaped and connected to physiologic monitoring devices during the visit
* Willingness to take amitriptyline daily for 8 weeks following study visit 1

Exclusion Criteria:

* Diagnosis of Crohn's disease, systemic sclerosis, known active ulcer disease, gastric cancer, or untreated/active Barrett's esophagitis based on subject self-report and/or medical record review
* Heavy alcohol use (> 6 drinks/week for women and > 13 drinks/week for men) based on subject self-report
* Pregnant, attempting to become pregnant, or breast-feeding
* Dementia or significant memory difficulties as determined by the study team and medical record review
* Severe, unstable psychiatric disease based on subject self-report, study team determination, and/or medical record review
* Bipolar disorder, concurrent treatment with a SSRI or another antidepressant that interacts with tricyclic antidepressants
* Prolonged QTc or severe heart disease
* History of seizure disorder
* Severe liver impairment - e.g., cirrhosis, hepatocellular carcinoma, hepatitis
* Currently taking a tricyclic antidepressant, allergy to tricyclic antidepressants, or another medical contraindication to taking amitriptyline or related medications
* Greater than 15 doses of nonsteroidal anti-inflammatory drugs (NSAIDS) within the prior 30 days (aspirin ≤ 325 mg daily permitted) or ongoing NSAID use at a level deemed likely to interfere with the study
* Failure to complete the baseline symptom diary for at least 6 of 7 days
* Change in GERD treatment regimen within the last 2 weeks (subjects may use antacids, H2 receptor blockers, and/or proton pump inhibitors as long as they are symptomatic on a stable regimen)
* Allergy to adhesives
* Inability to provide informed consent
* In the opinion of the investigator, unable to comply with the study protocol or has a condition that would likely interfere with the study

Ages: 24 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Dossett, MD, PhD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
Will need to request written permission and obtain a data sharing agreement and permission from the IRB to receive individual level participant data.

REFERENCES:
- [Background] Miner P Jr, Orr W, Filippone J, Jokubaitis L, Sloan S. Rabeprazole in nonerosive gastroesophageal reflux disease: a randomized placebo-controlled trial. Am J Gastroenterol. 2002 Jun;97(6):1332-9. doi: 10.1111/j.1572-0241.2002.05769.x. PMID 12094846
- [Background] Marci CD, Ham J, Moran E, Orr SP. Physiologic correlates of perceived therapist empathy and social-emotional process during psychotherapy. J Nerv Ment Dis. 2007 Feb;195(2):103-11. doi: 10.1097/01.nmd.0000253731.71025.fc. PMID 17299296

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Visit: A standardized visit (based on a pre-set question template) modeled after a primary care visit focused on evaluating GERD symptoms.
- Expanded Visit: A standardized visit (based on a pre-set question template) modeled after an integrative medicine visit for GERD symptoms. The Expanded Visit includes all of the questions in the Standard Visit plus additional questions about the nature of the GI symptoms (e.g., taste of reflux, food cravings and aversions), other health issues, and the patient's temperament (e.g., shy, anxious, caring). Some of these questions address the patient's "constitutional type" as might be assessed by some integrative practitioners (e.g., tell me about your sleep; do you tend to be hot or cold?).
Period: Overall Study
Arm/Group | Standard Visit | Expanded Visit
Started | 2 | 5
Completed | 2 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Visit | Expanded Visit | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (2.1) | 45.0 (16.0) | 45.4 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Average Daily GERD Symptom Severity [Mean (Standard Deviation); unit: units on a scale] — Severity of GERD symptoms were assessed by participant self-report on a 7-day symptom diary for one week immediately prior to enrolling in the study. Possible daily scores ranged from 0-12 with higher scores indicating more severe symptoms (sum of daytime heartburn, nighttime heartburn, and acid regurgitation symptoms each rated 0-4 in severity [none, mild, moderate, severe, very severe]). Daily values across each of the 7 days were averaged to create the average daily GERD symptom severity score.
  units on a scale | 2.9 (2.6) | 4.3 (4.6) | 3.9 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in GERD Symptoms
Description: Change in the average daily GERD symptom severity score over a 7-day period from baseline to the last week of the study in the expanded vs. standard group. GERD symptom severity is based on the sum of scores assessing the severity of daytime heartburn, nighttime heartburn, and acid reflux each on a 0-4 point scale (none, mild, moderate, severe, very severe; higher scores signify worse symptoms). Possible score range = 0 - 12. Change score calculated as average score at 8 weeks minus average score at baseline. For statistical testing, we used a general linear model of post-GERD symptoms adjusted for baseline GERD symptoms and randomization assignment.
Time Frame: Time 0 (baseline) to 8 weeks
Population: All enrolled participants who attended both baseline and 8 week follow-up visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Visit | Expanded Visit
Number analyzed (Participants) | 2 | 4
units on a scale | 0.6 (1.6) | -1.7 (3.7)
Statistical Analysis 1: Comparison: Standard Visit vs Expanded Visit; Test type: Superiority; p = 0.41, ANOVA

2. Secondary Outcome: Relationship of Physiologic Concordance in Skin Conductance Between Patient and Physician With Patients' GERD Symptom Change
Description: Concordance in skin conductance response (SCR) between patient and physician was calculated using an established approach to create a single index value for the visit (baseline). Average slopes of the SCR were calculated in moving 5 second windows, offset by 1 second. Pearson correlations between time-locked patient and physician SCR slopes were calculated over successive 15 second windows. A single session index was calculated from the ratio of the sum of the positive correlations across the entire visit divided by the sum of the absolute value of the negative correlations across the entire visit. To reduce skew, the natural logarithm of the index was calculated. An index value of zero reflects equal positive and negative correlations, a value greater than zero reflects more concordance in SCR than not, while a value less than zero reflects less than 50% concordance. In the statistical analysis, we included change in GERD symptoms from baseline to 8 weeks.
Time Frame: Time 0 (baseline) to 8 weeks.
Population: All enrolled participants with complete physiologic data for both the patient and physician.
Measure: Mean (Standard Deviation); unit: natural log of the index value
Arm/Group | Standard Visit | Expanded Visit
Number analyzed (Participants) | 2 | 4
natural log of the index value | 0.02 (0.47) | -2.2 (4.8)
Statistical Analysis 1: Comparison: Standard Visit vs Expanded Visit; For statistical testing, we used a general linear model of change in GERD symptoms from baseline to 8 weeks adjusted for the natural log of the index value (of the ratio of the change in skin conductance between patient and physician at baseline) and randomization assignment; Test type: Superiority; p = 0.09, ANOVA

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Standard Visit | Expanded Visit
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 0/2 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Visit (N=2) | Expanded Visit (N=5)
chest pain (Gastrointestinal disorders) | 0 | 1 — Secondary to GERD symptoms, resolved spontaneously. Not related to study interventions
Allergic reaction (Immune system disorders) | 0 | 1 — Developed an allergic reaction to a zio patch. Not related to study interventions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT04292470/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT04292470/ICF_001.pdf